CLINICAL TRIAL: NCT00769587
Title: Phase II Study of Thalidomide in Mastocytosis
Brief Title: Thalidomide in Treating Patients With Relapsed or Progressive Systemic Mastocytosis
Status: Completed | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI06-DR-DAMAJ; CHU-AMIENS-PI06; EUDRACT-2006-005087-10; INCA-RECF0510
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Non Neoplastic Condition; Precancerous Condition
Keywords: aggressive systemic mastocytosis; smoldering systemic mastocytosis
MeSH Terms: conditions — Precancerous Conditions; Mastocytosis, Systemic | interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Thalidomide (Experimental): Use of thalidomide
  Interventions: Drug: thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of systemic mastocytosis by blocking blood flow to the disease.

PURPOSE: This phase II trial is studying how well thalidomide works in treating patients with relapsed or progressive systemic mastocytosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the objective response rate at 6 months in patients with systemic mastocytosis treated with thalidomide.

Secondary

* Determine the tolerability of this drug in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral thalidomide once daily for 6 months in the absence of disease progression.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of systemic mastocytosis

  * Aggressive or borderline (smoldering) disease (in first line or more)
  * Relapsed or progressive disease
* Measurable or evaluable disease
* Presence of c-Kit D816V mutation in the skin, spine, or infiltrated organs
* No nonsymptomatic mastocytosis

PATIENT CHARACTERISTICS:

* Life expectancy > 3 months
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception for 1 month prior to, during, and until first menstrual cycle after completion of study treatment
* Bilirubin < 2 times normal (unrelated to disease)
* Liver enzymes < 2 times normal (unrelated to disease)
* Creatinine ≤ 300 mmol/L
* No central or peripheral neuropathy leading to psychiatric concerns
* No HIV positivity
* No active infection or other serious underlying illness that would preclude treatment
* No history of thromboembolism or deep vein thrombosis
* No geographical, social, or psychological reasons preventing medical monitoring

PRIOR CONCURRENT THERAPY:

* More than 4 weeks since prior antitumor therapy (e.g., chemotherapy, radiotherapy)
* No other concurrent treatment specific for this disease
* No concurrent participation in another experimental drug trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-06; Primary Completion 2011-05 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Objective reduction of the infiltration rate at 6 months | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Gandhi Damaj, Study Chair — Centre Hospitalier Universitaire, Amiens
Locations (1):
- Centre Hospitalier Universitaire d'Amiens, Amiens, France

REFERENCES:
- [Background] Gruson B, Lortholary O, Canioni D, Chandesris O, Lanternier F, Bruneau J, Grosbois B, Livideanu C, Larroche C, Durieu I, Barete S, Sevestre H, Diouf M, Chaby G, Marolleau JP, Dubreuil P, Hermine O, Damaj G. Thalidomide in systemic mastocytosis: results from an open-label, multicentre, phase II study. Br J Haematol. 2013 May;161(3):434-42. doi: 10.1111/bjh.12265. Epub 2013 Feb 22. PMID 23432617